CLINICAL TRIAL: NCT06610305
Title: Ovarian Hormone Withdrawal, Anhedonia, and Reward Sensitivity in Women With Premenstrual Exacerbations of Depression: A Crossover Randomized Controlled Trial
Brief Title: Ovarian Hormone Withdrawal, Anhedonia, and Reward Sensitivity in Women With Premenstrual Exacerbations of Depression
Acronym: PEAR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 24-1715; 1R01MH122446 (NIH)
Record Dates: First submitted 2024-09-17; First posted 2024-09-24 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder
Keywords: depression; hormone; premenstrual; estrogen; progesterone; perimenstrual
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Estradiol+Progesterone, then Placebo (Experimental): Two weeks of luteal phase transdermal estradiol (0.1mg/day)+oral progesterone (200 mg/day) during the first intervention cycle, followed by a one cycle washout, followed by two weeks of luteal phase transdermal/oral placebo
  Interventions: Drug: Transdermal estradiol; Drug: Progesterone; Drug: Transdermal placebo patch; Drug: placebo capsule
- Placebo, then Estradiol+Progesterone (Experimental): Two weeks of luteal phase transdermal/oral placebo during the first intervention cycle, followed by a one cycle washout, followed by two weeks of luteal phase transdermal estradiol (0.1 mg/day)+oral progesterone (200 mg/day)
  Interventions: Drug: Transdermal estradiol; Drug: Progesterone; Drug: Transdermal placebo patch; Drug: placebo capsule

INTERVENTIONS:
Drug: Transdermal estradiol — 0.1 mg/day delivered via weekly patch
Drug: Progesterone — 100 mg twice daily (200 mg/day total) administered via oral capsule
Drug: Transdermal placebo patch — Once weekly via transdermal patch
Drug: placebo capsule — Twice daily via oral capsule

SUMMARY:
The goal of this clinical trial is to learn how hormonal changes over the menstrual cycle affect mood symptoms in reproductive-aged women with depression that worsens during the premenstrual period. The main questions it aims to answer are:

--How do fluctuations in estradiol and progesterone across the menstrual cycle affect the ability to experience pleasure and the neural sensitivity to reward in hormone-sensitive, depressed women? And consequently, how does stabilizing the luteal phase decline in estrogen and progesterone (using estradiol patches and progesterone pills) affect these changes?

Participants will:

* Receive hormones followed by placebo, or vice versa, for a total of four weeks across three menstrual cycles
* Complete daily mood ratings
* Collect home urine samples for hormone testing
* Complete five biobehavioral testing sessions during which neural responses are recorded (via electroencephalography, or EEG) during an acute stress task and computer tasks

DETAILED DESCRIPTION:
Potential participants will first be screened over the phone to assess health history (including mental health) and reproductive status. Those who meet inclusion/exclusion criteria will be invited to an in-person enrollment session. At enrollment, consent will be obtained and participants will complete a structured interview and a series of questionnaires. Interested participants will be educated on the use of smartphone-based ecological momentary assessment (EMA) surveys, which will be used to complete daily mood ratings over the course of the study.

Following enrollment, women will complete daily mood ratings for one menstrual cycle using EMA; this is called the "prospective-assessment" phase. Those who meet our predetermined mood criteria during prospective assessment will move into a one-cycle lead-in phase of the study, where they will continue daily EMA; for those who do not, study participation will conclude. Participants will complete a single in-person visit during the lead-in phase, at which they will be randomized to one of two conditions within the randomized crossover design; they will also complete an acute stress task and computer tasks while EEG is recorded.

During the intervention phase, the first condition will receive transdermal estradiol (E2) (0.1mg/d)+oral progesterone (P4) (200mg/d) during the luteal phase of cycle 1 of the intervention phase (third cycle overall), and placebo (transdermal+oral) during the luteal phase of cycle 3 of the intervention phase (fifth cycle overall); the second will receive placebo during the luteal phase of intervention cycle 1, and transdermal E2+oral P4 during the luteal phase of intervention cycle 3. Cycle 2 will be a washout for both conditions (mood assessment only, without hormone collection or labs). During cycles 1 and 3, every-other-day urine samples will be collected for estradiol and progesterone metabolites and daily anhedonia symptoms will be assessed. Women will also complete two lab sessions tied to the mid-follicular and late luteal phases, as determined by a fixed time window relative to ovulation. At each lab session, EEG will be recorded during computer tasks that probe reward sensitivity, responses from which will serve as our primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Biologically female and between the ages of 18-45 years (45 set as upper limit to avoid endocrine changes associated with perimenopause).
* Self-reported regular menstrual cycles between 25 and 35 days.
* A previous diagnosis of major depressive disorder, with self-reported premenstrual worsening of symptoms.
* If the woman has children, she must be at least 1 year postpartum.
* English-speaking

Exclusion Criteria:

* Pregnant, breastfeeding, or trying to become pregnant. Pregnancy status will be confirmed using a urine pregnancy test at the enrollment visit and again at the first visit of the second condition. Women will be instructed to use a barrier method of birth control during the study.
* Taking any form of exogenous hormones or IUD, and must have ended previous use of hormonal preparations at least one month prior to the study. Women who were previously taking oral contraceptives or other hormonal medications must have one normal menstrual cycle (menstrual period) prior to enrollment in the study.
* BMI less than 18 or greater than 29.
* A personal history of any chronic medical condition that could confound the experimental protocol, including but not limited to metabolic or autoimmune disease, epilepsy, endometriosis, cancer, diabetes, cardiovascular, gastrointestinal, hepatic, renal, pulmonary disease, migraine with aura, hypertension, Parkinson's disease, chronic pain, and thromboembolic events.
* A family history indicative of increased risk of breast cancer or thromboembolic disorders.
* Current cigarette smoking.
* A history of mania, psychosis, or substance use disorder.
* Any recent history (last 12 months) of active suicidal ideation, or suicide attempt within the last 5 years.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Dimensional Anhedonia Rating Scale (Luteal Phase Stabilized vs Luteal Phase Unstabilized Hormones vs Follicular Phase) | 3 menstrual cycles (each cycle approximately 28 days in duration)
  Measures several domains of hedonic function, including desire, motivation, effort, and consummatory pleasure, across various contexts. 17 items, max score 68, higher scores indicate greater anhedonia.
Reward Positivity (Luteal Phase Stabilized vs Luteal Phase Unstabilized Hormones vs Follicular Phase) | Over the course of 2 menstrual cycles (~28 days each), EEG will be collected four times on four separate days: twice during the late luteal phase (11-14 days following ovulation), and twice during the mid follicular phase (23-25 days following ovulation)
  An EEG event-related potential reflecting sensitivity to positive feedback.

SECONDARY OUTCOMES:
Daily Record of Severity of Problems (Luteal Phase Stabilized vs Luteal Phase Unstabilized Hormones vs Follicular Phase) | 5 menstrual cycles (each cycle approximately 28 days in duration)
  Measures daily symptom burden used for the evaluation and diagnosis of menstrual-related mood disorders. The items measure symptoms related to core emotional disturbance, including depression, anxiety, irritability, and mood lability, as well as secondary symptoms such as concentration, energy, appetite, sleep, and physical symptoms and interference from symptoms overall. 24 items, scale range 24-144, higher scores indicate greater symptoms.
Inventory for Depression and Anxiety Symptoms (Luteal Phase Stabilized vs Luteal Phase Unstabilized Hormones vs Follicular Phase) | Over the course of 2 menstrual cycles (~28 days each), IDAS will be collected 4 times on 4 separate days: twice during the late luteal phase (11-14 days following ovulation), and twice during the mid follicular phase (23-25 days following ovulation)
  Measures depressive and anxiety symptoms within 10 different subdomains: Suicidality, Lassitude, Insomnia, Appetite Loss, Appetite Gain, Ill Temper, Well-Being, Panic, Social Anxiety, and Traumatic Intrusions. 64 items, scale range 64-320, higher scores indicate greater symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Chris Sikes-Keilp, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No